

### AIC316-03-I-01

# Summary of the Clinical Trial Protocol and Statistical Plan

A single-center, open-label, 2-period, fixed-sequence Phase 1 trial to evaluate the effect of esomeprazole on the pharmacokinetics of pritelivir

NCT number: NCT05513625

Investigational drug: Pritelivir

Sponsor: AiCuris Anti-infective Cures AG

Address: Friedrich-Ebert Str. 475

DE-42117 Wuppertal

Germany

Finalization dates:

Summary of the Clinical Trial 16Sep2022

Protocol and Statistical Plan, V1.0:

Clinical Trial Protocol, 04Jun2020

V1.0:

Safety Statistical Analysis Plan, 21Jul2020

V2.0:

Pharmacokinetic Statistical 01Jul2020

Analysis Plan, V1.0:

## Summary of the Clinical Trial Protocol and Statistical Plan

AIC316-03-I-01

V1.0 16Sep2022

## SUMMARY OF THE CLINICAL TRIAL PROTOCOL AND STATISTICAL PLAN

| Name of Sponsor/Company: | AiCuris Anti-infective Cures GmbH | |
|---|---|---|
| Title of the trial: A single-center, open-label, 2-period, fixed-sequence Phase 1 trial to evaluate the effect of esomeprazole on the pharmacokinetics of pritelivir | | |
| Principal Investigator: Dr. Leela Vrishabhendra | | |
| Trial center(s): | | |
| Medpace Clinical Pharmacology<br>5355 Medpace Way, Cincinnati, Ohio 45227, USA | | |
| Planned trial period: | | Phase of development: |
| First Subject First Visit:<br>Last Subject Last Visit | Jul 2020<br>Sep 2020 | Phase 1 |

#### **Objectives:**

- To investigate the effect of esomeprazole on the pharmacokinetics of pritelivir
- To investigate the pharmacokinetics of pritelivir metabolites AIC090015, AIC090105 and AIC090015-acylglucuronides
- To investigate the safety and tolerability of pritelivir

#### Trial design:

This will be a single-center, open-label, 2-period, fixed-sequence Phase 1 trial in 18 healthy adult male and female subjects (at least 7 subjects per sex). All subjects will receive treatment 1 (T1; single dose of 100 mg pritelivir will be administered on Day 1) in the first period, followed by treatment 2 (T2; single dose of 100 mg pritelivir will be administered on Day 1 and 40 mg esomeprazole will be administered qd from Day -3 to Day 1) in the second period. The wash-out period between pritelivir administrations in T1 and T2 is at least 4 weeks.

#### Number of subjects (planned):

1 8

#### Diagnosis and main criteria for inclusion:

Healthy adult male and female subjects (at least 7 subjects per sex) of any ethnic origin, aged 18 to 45 years inclusive.

#### Test product, dose and mode of administration:

Oral 100 mg pritelivir tablets

Oral 40 mg esomeprazole tablets (Nexium®)

#### **Duration of treatment:**

In Treatment Period 1:

Pritelivir: single dose of 100 mg on Day 1



### Summary of the Clinical Trial Protocol and Statistical Plan

AIC316-03-I-01

V1.0 16Sep2022

#### <u>In Treatment Period 2:</u>

4 days

Esomeprazole: 40 mg qd from Day -3 to Day 1, inclusive

Pritelivir: single dose of 100 mg on Day 1

#### Reference therapy, dose and mode of administration, batch number(s):

Not applicable.

Criteria for evaluation:

#### **Efficacy**

Not applicable.

#### **Pharmacokinetics**

#### Primary variables:

• AUC<sub>0-∞</sub>, AUC<sub>0-last</sub>, C<sub>max</sub> of pritelivir in plasma

#### Secondary variables:

- $t_{max}$ ,  $t_{lag}$ ,  $t_{1/2z}$ , CL/F,  $V_d$  /F, MRT of pritelivir in plasma
- AUC<sub>0-∞</sub>, AUC<sub>0-last</sub>, C<sub>max</sub>, t<sub>max</sub>, t<sub>lag</sub>, t<sub>1/2z</sub>, MRT of metabolites AIC090015, AIC090105 and AIC090015-acyl glucuronides in plasma
- The ratio between each of the metabolites AIC090015, AIC090105 and AIC090015-acyl glucuronides versus pritelivir will be calculated for AUC<sub>0-∞</sub>, AUC<sub>0-last</sub>

Pharmacokinetic profile will be determined in each period on Day 1 for 360 hours.

#### Pharmacogenomics/gene expression:

Post-hoc analysis of alleles associated with altered drug metabolism/ disposition may be determined.

#### **Safety**

- Overall tolerability
- Nature, frequency, duration, severity and causality of adverse events
- Clinical laboratory parameters
- Vital signs (blood pressure, pulse rate)
- Standard 12-lead ECG



### Summary of the Clinical Trial Protocol and Statistical Plan

AIC316-03-I-01

V1.0

16Sep2022

#### **Statistical methods:**

#### Pharmacokinetic data

The Pharmacokinetic Set (PKS) will include all subjects in the Safety Set (SS) with at least 1 plasma concentration time point for inclusion in the PK analysis. The PKS will be used for the PK analyses.

Descriptive statistics will be calculated for plasma concentrations of pritelivir and derived PK parameters. Statistics include sample size (n), mean, standard deviation (SD), %CV, geometric mean, median, minimum and maximum.

The relative bioavailability of pritelivir with respect to the primary variables  $AUC_{0-\infty}$ ,  $AUC_{0-last}$  and  $C_{max}$  will be explored based on the log transformed data with an analysis of variance model with treatment (as fixed effect) and subject (as random effect). Point estimates (GMR) and 90% confidence intervals (90% CIs) will be computed for the ratio T2 (test) /T1 (reference) to evaluate the effect of esomeprazole on pritelivir PK under fasted conditions.

#### Safety data

Safety data analysis will be conducted on the Safety Set. Statistical analysis of the safety data will be limited to descriptive summaries.

The results of AE recording, vital signs, 12-lead ECGs, clinical laboratory investigations, and physical examinations will be listed by subject and analyzed by descriptive statistics as appropriate.

All adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Incidences of treatment-emergent adverse events (TEAE) that began after the start of trial treatment (post-dose on Day 1 to End of trial examination) will be summarized at 3 levels: the overall subject level (occurrence of at least one TEAE), primary System Organ Class level, and preferred term level. All adverse events will be listed together with information on onset, duration, frequency, intensity, seriousness, relationship to IMP, outcome, and action taken.

Laboratory data will be presented in summary statistics of raw data and change from baseline values (mean, median, standard deviation, minimum, maximum), and by flagging values outside the reference range in data listings. Vital signs will be summarized presenting statistics of raw data and change from baseline values (mean, median, standard deviation, minimum and maximum).

ECG data will be summarized presenting statistics of raw data and change from baseline values (mean, median, standard deviation, minimum and maximum). In addition, 12-lead ECGs will be analyzed with a focus on the incidence and extent of QTc prolongation. QTc will be calculated according to Fridericia formula. Frequencies for classes of absolute values and differences from baseline will be provided according to the classifications defined by ICH-E14.

The World Health Organization Drug Dictionary (WHO-DD) will be used for coding of concomitant medications (except IMPs).